CLINICAL TRIAL: NCT01024933
Title: Trial Using Motivational Interviewing Positive Affect and Self-Affirmation in Hypertension (TRIUMPH)
Acronym: Triumph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Triumph; 1P60MD003421-01 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational and Behavioral (Placebo Comparator): The Education and Behavioral Contract (Control group) will receive an educational workbook and behavioral contract. Each patient will receive a home blood pressure device for self-monitoring, and will be called every two months.
  Interventions: Behavioral: Educational and Behavioral
- PASA group-intervention (Experimental): The PASA group (Positive Affect/Self-Affirmation/Motivational Interviewing) will receive a positive-affect and self-affirmation intervention with motivational interviewing.These patients will also receive an educational workbook and behavioral contract. This is the intervention.
  Interventions: Behavioral: Positive Affect/Self-Affirmation/Motivational Interviewing

INTERVENTIONS:
Behavioral: Positive Affect/Self-Affirmation/Motivational Interviewing — The PASA group-intervention will receive small gifts one week prior to their scheduled follow up. The PASA intervention involves reminding participants to think about their proud and positive moments. The motivational interviewing intervention includes assessing the patient's motivation and confidence; elicit barriers and concerns; summarize in a non-threatening manner the 'pros' and 'cons' of patient's concerns, thereby eliciting positive self-motivational statements about the behavior. Follow up will be every two months.
  Arms: PASA group-intervention
Behavioral: Educational and Behavioral — The Education and Behavioral Contract (Control group)will receive an educational workbook and behavioral contract. In addition, each patient will receive a home blood pressure device for self-monitoring, and will be called every two months.
  Arms: Educational and Behavioral

SUMMARY:
The primary aim of this study is to evaluate whether an intervention that combines positive affect and self-affirmation with motivational interviewing (TRIUMPH) improves blood pressure control compared to an educational/behavioral contract intervention at 12 months. We hypothesize that a greater proportion of participants in the experimental arm of TRIUMPH will have adequate blood pressure control as defined by Seventh Joint National Committee on Detection, Evaluation and Treatment of Hypertension (JNC-7.)

DETAILED DESCRIPTION:
TRIUMPH is designed to build on the findings of our previous studies by combining positive affect and self affirmation with motivational interviewing in order to increase blood pressure control in community based practices that care for large numbers of hypertensive black patients. Patients in both the educational and behavioral contract control group and would receive a workbook, would make a behavioral contract, and a home blood pressure monitor. The positive affect/self-affirmation group would receive the same components as the control group. In addition the experimental group would receive a positive affect/self-affirmation induction and motivational interviewing.

Both the control group and the experimental group would be followed at 2 month intervals. The outcome blood pressure control in this group will be contrasted to the knowledge/behavioral contract group. We hypothesize that we can increase the percent of patients who have blood pressure control to 75%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Must be receiving care within the Renaissance Health Network for at least one year.
* Must have uncontrolled HTN defined as an average SBP>140 mmHg or DBP>90 mmHg on at least two previous visits in the past year and be taking at least one antihypertensive medication.
* Must self-identify as Black, or African American.
* Must have patient's physician to participate in the study.

Exclusion Criteria:

* Being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that he/she could not complete all requested tasks).
* Participation in other clinical trials.
* Diagnosis of cognitive dysfunction or significant psychiatric comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the blood pressure control. | 12 months

SECONDARY OUTCOMES:
The secondary outcome is within-patient change in Systolic Blood Pressure and Diastolic Blood Pressure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Lincoln Medical and Mental Health Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share